CLINICAL TRIAL: NCT03034889
Title: Neurocognitive Development in Children Who Received General Anesthesia Before the Age of 3 Years: A Historic-prospective, Controlled, Single Center Cross-section Trial
Brief Title: Anesthesia Related Neurocognitive Deficits in Children
Acronym: ANFOLKI-36
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Tino Münster, Prof. Dr., University of Erlangen-Nürnberg Medical School
Other Study IDs: ANFOLKI-36
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia
Keywords: Anesthesia; Children; General Anesthesia; Neurocognitive Outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: Children age 4-10 who required general anesthesia before the age of 36 months in the context of surgical and diagnostic procedures or sedation during intensive care, excluding neurosurgical interventions or cardiac surgery as well as preexisting hereditary or acquired neurocognitive deficits
- Control: Children age 4-10 who did not require any anesthesia before the age of 36 months. Excluding preexisting hereditary or acquired neurocognitive deficits.

SUMMARY:
The infantile brain has to pass essential, mayor steps in the first 36 months of life. During that period of development it is particularly vulnerable to toxic, exogenic influences. This study wants to review the long-term effects of children who were exposed to anesthesia in the first three years of their life. Therefore the investigators will examine children at age of 4-10 that were exposed to anesthesia and compare their neurocognitive capacity to children who did not have any exposure to anesthesia. The investigators plan on measuring the intelligence quotient using standardized tests which will be performed by a trained psychologist. In addition there will be a questionnaire concerning behavioral characteristics and educational development which is filled by the parents. The exposed children will be recruited from our preexisting database, the control group will be recruited from practitioners and the pediatric walk-in-clinic.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia before the age of 36 months

Exclusion Criteria:

* neurosurgical interventions
* cardiac surgery
* preexisting hereditary or acquired cognitive deficits
* no informed consent

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children age 4-10 who underwent general anesthesia below the age of 36 months in context of surgical or diagnostic procedures or sedation uring intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Capacity for children between 7 and 10 years of age | Test is done 1 to 10 years after anesthesia and is lasting 3 hours
  Standardized tests for intelligence quotient (IQ): Kaufman Assessment Battery for Children - Second Edition (KABC-II)
Cognitive Capacity for children between 4 and 7 years of age | Test is done 1 to 10 years after anesthesia and is lasting 3 hours
  Standardized tests for intelligence quotient (IQ): Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III)
Cognitive Capacity for children between 2 and 4 years of age | Test is done 1 to 10 years after anesthesia and is lasting 3 hours
  Standardized tests for intelligence quotient (IQ): Wechsler Intelligence Scale for Children (WISC-IV)

SECONDARY OUTCOMES:
Educational status | 1 to 10 years after anesthesia, lasting 30 minutes
  Questionnaire, filled by parents 1-10 years after anesthesia exposure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Erlangen, Bavaria, Germany